CLINICAL TRIAL: NCT01662921
Title: Non-inferiority Trial Comparing Insulin Glulisine to Insulin Lispro as Part of a Basal-bolus Insulin Regimen for the Treatment of Gestational Diabetes.
Brief Title: Comparator Trial Using Insulin Glulisine vs. Insulin Lispro for Treatment of Gestational Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sansum Diabetes Research Institute (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APIDRL06229
Record Dates: First submitted 2012-08-07; First posted 2012-08-13 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Diabetes During Pregnancy
Keywords: bolus treatment
MeSH Terms: conditions — Diabetes, Gestational | interventions — Isophane Insulin, Human; Insulin Lispro; insulin glulisine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NPH and insulin lispro (Active Comparator): Patients diagnosed with diabetes during pregnancy will be randomized to long acting insulin NPH and short acting insulin lispro in a basal bolus regimen to treat post prandial hyperglycemia using a dosing schedule of 50% NPH calculated by the patients weight and gestational age and 50% lispro pending their last three SMPG average.
  Interventions: Drug: NPH; Drug: Insulin LISPRO
- NPH and insulin glulisine (Active Comparator): Patients with a diagnosis of diabetes during pregnancy will be randomized to using long acting insulin NPH and short acting insulin glulisine as treatment for post prandial hyperglycemia with a 50% NPH dosing schedule based on the weight and gestational age and 50% glulisine schedule based on their last three SMBG result average.
  Interventions: Drug: NPH; Drug: Insulin glulisine

INTERVENTIONS:
Drug: NPH — Long acting insulin NPH dosing will be titrated weekly derived from the patients current weight and gestational age
  Other Names: Humulin N, Novolin N
Drug: Insulin LISPRO — Insulin lispro dosing will be titrated weekly based on the patient's average SMBG readings from each meal during the past three days
  Other Names: Humalog
  Arms: NPH and insulin lispro
Drug: Insulin glulisine — Insulin glulisine will be titrated weekly based on the patient's average SMBG readings from each meal during the past three days
  Other Names: Apidra
  Arms: NPH and insulin glulisine

SUMMARY:
We hypothesize that insulin glulisine is non-inferior to currently proven rapid-acting insulin lispro when used in a basal/bolus regimen to treat hyperglycemia in patients with gestational diabetes mellitus.

DETAILED DESCRIPTION:
To date, only two rapid-acting insulin analogs have been shown to be safe and effective for the treatment of diabetes during pregnancy: insulin aspart and insulin lispro.

The pharmacokinetics and pharmacodynamics of insulin glulisine are unique and insulin glulisine may be the best rapid-acting analog for the treatment of post-prandial hyperglycemia. We believe that insulin glulisine should be evaluated in women with gestational diabetes for its potential efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent to participate in clinical trial
* Pregnant and 20-30 weeks gestation
* Diagnosed with gestational diabetes
* Failed diet therapy (failed lifestyle modification will be defined as 10% or greater SMBG values above pre-meal <90mg/dL and post prandial < 120mg/dL
* Eat at least 2 meals per day

Exclusion Criteria:

* Pregnant women <18 years old
* Blood pressure > 140/80 mmHg
* A1C equal to or greater than 6.5% at time of enrollment
* Pre-pregnancy BMI > 40Kg/m squared
* Evidence of any fetal anomaly on any fetal ultrasound
* Currently using hypoglycemic agent
* Refusal to use insulin before meals
* Inability to understand instructions or to consent to participate
* Pregnant women with history of T1DM or T2DM
* Clinical judgment by investigator that patient is inappropriate for clinical trial or has a metabolic disorder that could interfere with results

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2015-01-31 (Actual); Study Completion 2015-08-31 (Actual)

PRIMARY OUTCOMES:
show that insulin glulisine is non-inferior to insulin lispro in a basal/bolus regimen to treat hyperglycemia in patient with gestational diabetes mellitus | week 4 of insulin treatment
  compare average 1-hour post prandial SMBG measurements between patients randomized to insulin glulisine or insulin lispro

SECONDARY OUTCOMES:
Serum blood glucose area under the curve (AUC) at one 4-hour in-clinic meal challenge | week 2 of insulin treatment
  patients will come to the study site under fasting conditions and eat a standardized meal in the morning post administration of insulin NPH and their randomized bolus insulin.
Compare A1C at enrollment and weekly until delivery | up to 36 weeks
  A1C is measured weekly at each pregnancy visit up to 26 visits. Subjects are enrolled at 20-32 weeks gestation and have weekly visits to obtain A1C through delivery, and again at the 6-week postpartum visit.
Compare incidence of hypoglycemic episodes <60 mg/dL with symptoms | up to 36 weeks
  Hypoglycemic episodes since the last visit will be reported at each pregnancy visit, usually weekly, from enrollment at 10-30 weeks gestation through delivery and at the 6-week postpartum visit if continuing to take insulin.

OTHER OUTCOMES:
Compare incidence of birth weight >90th percentile | delivery
Compare incidence of primary cesarean section | delivery

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Castorino, DO, Principal Investigator — Sansum Diabetes Research Institute; Leonie Mattison, PhD, Study Director — Sansum Diabetes Research Institute
Locations (1):
- William Sansum Diabetes Center, Santa Barbara, California, United States

REFERENCES:
- [Background] 1. Centers for Disease Control and Prevention: National diabetes fact sheet: national estimates and general information on diabetes and prediabetes in the United States, 2011. Atlanta, GA: U.S. Department of Health and Human Services, Centers for Disease Control and Prevention, 2011.
- [Background] Castorino K, Jovanovic L. Pregnancy and diabetes management: advances and controversies. Clin Chem. 2011 Feb;57(2):221-30. doi: 10.1373/clinchem.2010.155382. Epub 2010 Dec 9. PMID 21148303
- [Background] HAPO Study Cooperative Research Group; Metzger BE, Lowe LP, Dyer AR, Trimble ER, Chaovarindr U, Coustan DR, Hadden DR, McCance DR, Hod M, McIntyre HD, Oats JJ, Persson B, Rogers MS, Sacks DA. Hyperglycemia and adverse pregnancy outcomes. N Engl J Med. 2008 May 8;358(19):1991-2002. doi: 10.1056/NEJMoa0707943. PMID 18463375
- [Background] Jovanovic L, Pettitt DJ. Treatment with insulin and its analogs in pregnancies complicated by diabetes. Diabetes Care. 2007 Jul;30 Suppl 2:S220-4. doi: 10.2337/dc07-s220. No abstract available. PMID 17596476
- [Background] Arnolds S, Rave K, Hovelmann U, Fischer A, Sert-Langeron C, Heise T. Insulin glulisine has a faster onset of action compared with insulin aspart in healthy volunteers. Exp Clin Endocrinol Diabetes. 2010 Oct;118(9):662-4. doi: 10.1055/s-0030-1252067. Epub 2010 Apr 28. PMID 20429049
- [Background] Manderson JG, Patterson CC, Hadden DR, Traub AI, Ennis C, McCance DR. Preprandial versus postprandial blood glucose monitoring in type 1 diabetic pregnancy: a randomized controlled clinical trial. Am J Obstet Gynecol. 2003 Aug;189(2):507-12. doi: 10.1067/s0002-9378(03)00497-6. PMID 14520226
- See also: Web page for Sansum Diabetes Research Institute — http://www.sansum.org